CLINICAL TRIAL: NCT04446637
Title: Comparison of Acute Bronchodilator Effects of Ipratropium/Levosalbutamol 20/50 mcg Fixed Dose Combination Delivered Via pMDI and Salbutamol 100 mcg Inhaler Plus Ipratropium 20 mcg Inhalation Aerosol in Patients With Stable Moderate-Severe-Very Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Acute Bronchodilator Effects of Ipratropium/Levosalbutamol 20/50 mcg Fixed Dose Combination vs Salbutamol 100 mcg Inhaler Plus Ipratropium 20 mcg Inhalation Aerosol Free Combination in Patients With Stable COPD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: administrative decision
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-01.19
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, ipratropium, levosalbutamol, levalbuterol, salbutamol, albuterol, MDI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Albuterol; Suspensions; Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: Multicenter, single day, noninferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipratropium/Levosalbutamol (Experimental): Ipratropium/Levosalbutamol 20/50 mcg Fixed Dose Combination (2 inhalations) via pMDI
  Interventions: Drug: Ipratropium/Levosalbutamol 20/50 mcg Fixed Dose Combination (2 inhalations) via pMDI
- Salbutamol + Ipratropium (Active Comparator): Salbutamol 100 mcg Inhaler (2 inhalations) + Ipratropium 20 mcg Inhalation Aerosol (2 inhalations) Free Combination via MDI
  Interventions: Drug: Salbutamol 100 mcg Inhaler (2 inhalations) + Ipratropium 20 mcg Inhalation Aerosol (2 inhalations) Free Combination via MDI

INTERVENTIONS:
Drug: Ipratropium/Levosalbutamol 20/50 mcg Fixed Dose Combination (2 inhalations) via pMDI — Ipratropium/Levosalbutamol 20 mcg/50 mcg Aerosol Inhalation, Suspension 2 inhalations in the morning (single day)
  Other Names: IPRALEV 20 mcg/50 mcg Aerosol Inhalation, Suspension
  Arms: Ipratropium/Levosalbutamol
Drug: Salbutamol 100 mcg Inhaler (2 inhalations) + Ipratropium 20 mcg Inhalation Aerosol (2 inhalations) Free Combination via MDI — Salbutamol 100 mcg Inhaler, 2 inhalations + Ipratropium 20 mcg Inhalation Aerosol,2 inhalations in the morning (single day).
  Other Names: VENTOLİN İnhaler 100 mcg + ATROVENT N MDI 0,02 mg/dose
  Arms: Salbutamol + Ipratropium

SUMMARY:
The purpose of this study is to compare acute bronchodilator effects of Ipratropium/Levosalbutamol 20/50 mcg Fixed Dose Combination (2 inhalations) via pMDI and Salbutamol 100 mcg Inhaler (2 inhalations) plus Ipratropium 20 mcg Inhalation Aerosol (2 inhalations) Free Combination in Patients with stable moderate-severe-very severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged ≥40 years diagnosed with symptomathic stable moderate-severe-very severe COPD: post-bronchodilator FEV1/FVC <70% predicted and a post-bronchodilator FEV1 <80% predicted at screen visit.

Group B COPD CAT: ≥10 or mMRC: ≥ 2 Exacerbation: 0-1 (not leading to hospital admission)

Group C COPD CAT: <10 or mMRC: 0-1 Exacerbation: ≥2 (not leading to hospital admission) or ≥1 (leading to hospital admission)

Group D COPD CAT: ≥10 or mMRC: ≥ 2 Exacerbation: ≥2 (not leading to hospital admission) or ≥1 (leading to hospital admission)

* Current or ex-smokers with a smoking history of at least 10 pack-years
* Patients who have no exacerbation within the last 4 weeks
* Female patients who use effective contraception
* Patients who have a capability to communicate with investigator
* Patients who accept to comply with the protocol
* Patients who sign written informed consent form

Exclusion Criteria:

* History of hypersensitive to anticholinergics or SABAs
* History of COPD exacerbation or lower respiratory track infection that required treatment with antibiotic, oral or parenteral corticosteroid within the last 4 weeks prior the screening visit or during the run-in/wash-out period or history of respiratory tract infection that required treatment with antibiotic within the last 14 days prior the screening visit.
* Hospitalization due to COPD or pneumonia within the last 3 mounts prior the screening visit
* Use of oral corticosteroid at unstable dosages (i.e. <6 weeks on a stable dose of prednisone)
* SGOT (serum glutamic oxaloacetic transaminase) >80 IU/L, SGPT (serum glutamic pyruvic transaminase) >80 IU/L, bilirubin >2.0 mg/dL or creatinine >2.0 mg/dL
* History of asthma, significant chronic respiratory diseases (i.e., significant bronchiectasis, interstitial lung diseases, etc.) other than COPD or presence of disease that may be serious and/or potentially affect results of the study.
* Initiation of an inhaled steroid or change in dose within <6 weeks prior the screening visit
* Use of beta-blocker, monoamine oxidase (MAO) inhibitor or tricyclic antidepressant within the last 30 days prior the screening visit
* Recent (within ≤1 year prior the screening visit) history of heart attack, heart failure, acute ischemic heart disease or presence of serious cardiac arrhythmia requiring drug treatment
* Regularly use of daytime CPAP (continuous positive airway measure) oxygen therapy for longer than 1 hour per day
* Initiation of pulmonary rehabilitation within the 3 months prior the screening visit
* History of lung volume reduction surgery
* Drug or alcohol abuse
* Presence of active tuberculosis
* History of atopy or allergic rhinitis
* History of cancer within the last 5 years
* Attenuated live virus vaccination within the last 2 weeks prior the screening visit or during the run-in/wash-out period
* Pregnancy or lactation
* Presence of known symptomatic prostatic hypertrophy requiring treatment
* Presence of known narrow-angle glaucoma requiring treatment
* Currently participating in another clinical trial or treatment with another investigational study drug within the last month or 6-half-lives, whichever is longer.

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-03 (Estimated); Primary Completion 2022-09-03 (Estimated); Study Completion 2022-09-03 (Estimated)

PRIMARY OUTCOMES:
FEV1 AUC (0-8h) | Baseline, 0 to 8 hours post-dose at treatment day
  Change From Baseline in Forced Expiratory Volume in one second (FEV1) Area Under the Curve (AUC) 0-8h.
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.

SECONDARY OUTCOMES:
FEV1 AUC (0-4h) | Baseline, 0 to 4 hours post-dose at treatment day
  Change From Baseline in FEV1 AUC (0-4h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
FEV1 AUC (4-6h) | Baseline, 4 to 6 hours post-dose at treatment day
  Change From Baseline in FEV1 AUC (4-6h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
FEV1 AUC (6-8h) | Baseline, 6 to 8 hours post-dose at treatment day
  Change From Baseline in FEV1 AUC (6-8h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
FVC AUC (0-4h) | Baseline, 0 to 4 hours post-dose at treatment day
  Change From Baseline in Forced Vital Capacity (FVC) AUC (0-4h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
FVC AUC (4-6h) | Baseline, 4 to 6 hours post-dose at treatment day
  Change From Baseline in FVC AUC (4-6h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
FVC AUC (6-8h) | Baseline, 6 to 8 hours post-dose at treatment day
  Change From Baseline in FVC AUC (6-8h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
FVC AUC (0-8h) | Baseline, 0 to 8 hours post-dose at treatment day
  Change From Baseline in FVC AUC (0-8h). Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
Change From Baseline in FEV1 and FVC within the first 15 minutes after dosing | Baseline, 0 to 15 minutes post-dose at treatment day
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
Mean Maximum Change From Baseline in FEV1 and FVC within the first 2 hours after dosing | Baseline, 0 to 2 hours post-dose at treatment day
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
Mean Maximum Change From Baseline in FEV1 and FVC over a period of 8 hours | Baseline, 0 to 8 hours post-dose at treatment day
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
The Time to Onset of Bronchodilator Response | Baseline, 0 to 8 hours post-dose at treatment day
  Bronchodilator response is defined as 100 mL improvement in FEV1. Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
The Time to Maximum Effect | Baseline, 0 to 8 hours post-dose at treatment day
  Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
Duration of Bronchodilator Response | Baseline, 0 to 8 hours post-dose at treatment day
  Bronchodilator response is defined as 100 mL improvement in FEV1. Spirometric measurements will be performed pre-treatment and 5 min, 15 min, 30 min, 45 min and 1 h, 2 h, 3 h, 4 h, 5 h, 6h, 7h, 8h after drug administration.
Evaluation of Safety (physical examination, numbers of adverse reactions and abnormal laboratory values or ECG related to treatment) | Baseline, 0 to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Hanta, Professor Doctor, Principal Investigator — Cukurova University Faculty of Medicine, Chest Diseases Department Adana - Turkey; Hakan Gunen, Professor Doctor, Principal Investigator — Sureyyapasa Training and Research Center for Chest Diseases and Thoracic Surgery, Maltepe, Istanbul - Turkey

IPD SHARING:
Plan to Share IPD: No